CLINICAL TRIAL: NCT05996757
Title: Effect of Wet Clothing Removal in the Treatment of Accidental Hypothermia: A Human Crossover Field Study
Brief Title: Effect of Wet Clothing Removal Compared to Use of a Vapor Barrier in Accidental Hypothermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/150
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Accidental Hypothermia; Emergencies
Keywords: Accidental hypothermia; Mountain Medicine
MeSH Terms: conditions — Hypothermia; Emergencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wet clothing removal (Active Comparator)
  Interventions: Procedure: Wet clothing removal
- Vapor barrier (No Intervention)

INTERVENTIONS:
Procedure: Wet clothing removal — The participants in the intervention group will have their clothing removed prior to insulation.
  Arms: Wet clothing removal

SUMMARY:
The optimal method of prehospital insulation and rewarming of hypothermic patients have been subject of debate, and there is a substantial lack og high-quality evidence to guide providers.

One question concerns whether or not the patients clothing should be removed prior to being wrapped in an insulating model with a vapor barrier. Evaporative heat loss is one of four mechanisms of heat loss, and preventing evaporative heat loss should be a prioritized task for providers. Removal of wet clothing usually means subjecting the patient to the environment, but will reduce the evaporative heat loss considerably. An other alternative is to encapsulate the patient in a vapor barrier. Evaporative heat loss will stop when the humidity inside the vapor barrier reaches 100%.

We aim to investigate whether it is recommended to removed wet clothing or encase the patient in a vapor barrier.

ELIGIBILITY:
Inclusion Criteria:

* Age <18
* American Society of Anaesthesiologists class 1
* No nicotine use

Exclusion Criteria:

* Acute illness on study day, fever or malaise

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2017-03-21 (Actual)

PRIMARY OUTCOMES:
Mean skin temperature | 60 minutes
  Change in mean skin temperature during rewarming phase

SECONDARY OUTCOMES:
Subjective thermal comfort and shivering | 60 minutes
  Using a validated questionnaire at regular intervals

CONTACTS AND LOCATIONS:
Overall Officials: Øyvind Thomassen, MD, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Henriksson O, Lundgren PJ, Kuklane K, Holmer I, Giesbrecht GG, Naredi P, Bjornstig U. Protection against cold in prehospital care: wet clothing removal or addition of a vapor barrier. Wilderness Environ Med. 2015 Mar;26(1):11-20. doi: 10.1016/j.wem.2014.07.001. PMID 25712295
- [Derived] Hagen LT, Brattebo G, Dipl-Math JA, Wiggen O, Osteras O, Mydske S, Thomassen O. Effect of wet clothing removal on skin temperature in subjects exposed to cold and wrapped in a vapor barrier: a human, randomized, crossover field study. BMC Emerg Med. 2024 Jan 25;24(1):18. doi: 10.1186/s12873-024-00937-8. PMID 38273259